CLINICAL TRIAL: NCT01404897
Title: Effects of a Modified Lower Carbohydrate, Higher Fat DASH Diet Plan on Plasma Lipids, Lipoprotein Particle Size, and Blood Pressure in Healthy Adults
Brief Title: Effects of High Fruit, Vegetable, and Dairy Intake on Plasma Lipids and Blood Pressure in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MM3274
Record Dates: First submitted 2011-07-22; First posted 2011-07-28 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Cardiovascular Disease; Dyslipidemia; Blood Pressure
Keywords: carbohydrate; DASH diet; blood pressure; cholesterol
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary Intervention: Control Diet (Experimental)
  Interventions: Other: Dietary Intervention
- Dietary Intervention: DASH-based diet (Experimental)
  Interventions: Other: Dietary Intervention
- Dietary Intervention: Modified DASH diet (Experimental)
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — 3 weeks of a typical Western diet pattern. 48% carbohydrate, 15% protein, 37% fat.
  Arms: Dietary Intervention: Control Diet
Other: Dietary Intervention — 3 weeks of a diet based on the Dietary Approaches to Stop Hypertension (DASH) diet plan. 57% carbohydrate, 18% protein, 25% fat.
  Arms: Dietary Intervention: DASH-based diet
Other: Dietary Intervention — 3 weeks of a reduced carbohydrate, higher fat modification of the DASH diet plan. 42% carbohydrate, 18% protein, 40% fat.
  Arms: Dietary Intervention: Modified DASH diet

SUMMARY:
The Dietary Approaches to Stop Hypertension (DASH) trial has been shown to reduce blood pressure and plasma total and LDL-cholesterol (C) compared to a Western diet, but shows no benefit on other blood lipid variables associated with cardiovascular disease (CVD) risk, namely HDL-cholesterol and triglycerides. The overall objective of this study is to determine whether modification of the DASH diet by substituting carbohydrate with fat will result in improvements in multiple biomarkers of CVD risk. Specifically, the investigators will test the hypotheses that modification of the DASH diet by reducing carbohydrate, primarily in the form of simple sugars and glycemic starches, and allowing for a more liberal intake of total and saturated fat, primarily from dairy foods, will: (1) improve lipoprotein markers of CVD risk (reduced total/HDL-C ratio, apolipoprotein B, small LDL particles, and increased HDL-C, apoAI, and large HDL particles); and (2) result in comparable reductions of systolic and diastolic blood pressure to those achieved with the standard DASH diet. The investigators will also assess the effects of the modified DASH diet on markers of insulin resistance and inflammation. Our main hypotheses will be tested by a controlled dietary intervention conducted in 40 healthy men and women who will be randomly allocated to consume, for 3 weeks each, a control Western diet, a standard DASH diet, and a modified low-carbohydrate DASH diet, separated by 2-week washout periods.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 years and older
* Average systolic blood pressure <160 mm Hg and diastolic blood pressure 80 - 95 mm Hg measured on 2 separate days
* Non-smoking
* Agrees to abstain from alcohol and dietary supplements during the study
* Willing to consume all study foods as instructed

Exclusion Criteria:

* History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, diabetes, lung disease, HIV, or cancer (other than skin cancer) in the last 5 years.
* Taking hormones or drugs known to affect lipid metabolism or blood pressure.
* Body Mass Index (BMI) > 35
* Total- and LDL-cholesterol > 95th percentile for sex and age.
* Fasting triglycerides > 500 mg/dl.
* Fasting blood sugar (FBS) > 126 mg/dl.
* Abnormal thyroid stimulating hormone
* Not weight stable
* Pregnant or breast-feeding

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total:HDL-cholesterol ratio | 4 weeks
HDL-cholesterol | 4 weeks
Apolipoprotein B | 4 weeks
Apolipoprotein AI | 4 weeks
Small LDL particles | 4 weeks
Large HDL particles | 4 weeks
Total:HDL-cholesterol ratio | 9 weeks
Total:HDL-cholesterol ratio | 14 weeks
HDL-cholesterol | 9 weeks
HDL-cholesterol | 14 weeks
Apolipoprotein B | 9 weeks
Apolipoprotein B | 14 weeks
Apolipoprotein AI | 9 weeks
Apolipoprotein AI | 14 weeks
Small LDL particles | 9 weeks
Small LDL particles | 14 weeks
Large HDL particles | 9 weeks
Large HDL particles | 14 weeks

SECONDARY OUTCOMES:
Blood Pressure | End of each experimental diet (4 wks, 9 wks, and 14 wks)
Triglycerides | End of each experimental diet (4 wks, 9 wks, and 14 wks)
Total Cholesterol | End of each experimental diet (4 wks, 9 wks, and 14 wks)
LDL-Cholesterol | End of each experimental diet (4 wks, 9 wks, and 14 wks)
Lipoprotein Subclasses (HDL, LDL, IDL, VLDL) | End of each experimental diet (4 wks, 9 wks, and 14 wks)
HOMA-IR | End of each experimental diet (4 wks, 9 wks, and 14 wks)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Children's Hospital Oakland Research Institute, Berkeley, California, United States

REFERENCES:
- [Derived] Chiu S, Bergeron N, Williams PT, Bray GA, Sutherland B, Krauss RM. Comparison of the DASH (Dietary Approaches to Stop Hypertension) diet and a higher-fat DASH diet on blood pressure and lipids and lipoproteins: a randomized controlled trial. Am J Clin Nutr. 2016 Feb;103(2):341-7. doi: 10.3945/ajcn.115.123281. Epub 2015 Dec 30. PMID 26718414